CLINICAL TRIAL: NCT01418066
Title: Feasibility and Safety of Ayurvedic Herbs in Diarrhoea-predominant Irritable Bowel Syndrome
Brief Title: Ayurvedic Herbs in Diarrhea Predominant Irritable Bowel Syndrome
Acronym: AHIB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Jost Langhorst, Prof. Dr., Universität Duisburg-Essen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-4673 AHIB
Record Dates: First submitted 2011-08-15; First posted 2011-08-16 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Tea decoction made of Graminis Flores abd Maidis stigmata.
  Interventions: Drug: Placebo tea
- Ayurvedic herbs (Experimental): Tea decoction made of Murraya koenigii leaves, Punica granatum and Curcuma
  Interventions: Drug: Ayurvedic Herbs

INTERVENTIONS:
Drug: Ayurvedic Herbs — A tea made of Murraya koenigii leaves, Punica granatum and Curcuma as powder. Decoction of 12ml powder in 100ml hot water is taken twice daily at least 30 minutes before a meal.
  Arms: Ayurvedic herbs
Drug: Placebo tea — Graminis Flores and Maidis stigmata as a powder. Decoction made of 12ml in 100ml hot water. To drink twice daily at least 30 Minutes before a meal.
  Arms: Placebo

SUMMARY:
In the present study the investigators are trying to evaluate the effect of Murraya koenigii leaves, Punica granatum and Curcuma which is administered to the patients in a combined form as tea. This study will help to evaluate the effect of these preparations scientifically in improving the IBS symptoms.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* Irritable Bowel Syndrome according to Rom-III
* Subtype Diarrhea or Alternating
* discomfort or pain > 1 times a week
* discomfort or pain > 4 on a Visual Analog Scale

Exclusion Criteria:

* Inflammatory bowel diseases (test results necessary)
* Lactose, Fructose Malabsorption (test results necessary)
* Celiac Disease
* Pregnancy or Breastfeeding
* Colectomy or Hemicolectomy >50cm
* Severe metabolic disorders, hormonal disorders, cardiac or respiratory failure, liver or renal diseases
* severe depression, psychotic or psychiatric disorders, substance abuse
* cancer within the last 5 years
* allergy to caraway
* acute inflammatory diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
irritable bowel syndrome- symptom severity score | T2 (Day 28)
  IBS-SSS(Francis, 1997)

SECONDARY OUTCOMES:
Frequency of abdominal discomfort/Pain | last week of treatment (days 21-28)
  Diary, daily rating of pain
Intensity of Abdominal Pain/Discomfort | Last week of treatment (days 21-28)
  Diary, daily rating of pain on a 100mm Visual Analog Scale
Stool and diarrhea Frequency | last week of treatment (days 21-28)
  Diary, daily counts
Quality of life | T2 (Day 28)
  measured with the EQ-5D
IBS Specific Quality of life | T2 (Day 28)
  measured with the IBS-QOL (Patrick, 1998)
Depression and Anxiety | T2 (day 28)
  HADS questionnaire (Hermann, 1995)
Adequate Relief Score | at day 7, 14, 21 and 28
  Adequate Relief Score (Mangel, 1998)
Global improvement | at days 7, 14, 21 and 28
  Question on global improvement: How have your symptomes changed compared to the last week: from much worse to much better on a 7-point scale
adverse events | up to week 15
  all adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jost Langhorst, Prof., MD, Principal Investigator — University Duisburg-Essen, Chair of Integrative Gastroenterology
Locations (1):
- Klinik für Naturheilkunde und Integrative Medizin, Essen, North Rhine-Westphalia, Germany